CLINICAL TRIAL: NCT00214656
Title: "Salvage Use" of Recombinant Activated Factor VII After Inadequate Haemostatic Response to Conventional Therapy in Complex Cardiac Surgery - a Randomised Placebo Controlled Trial
Brief Title: "Salvage Use" of Recombinant Factor VIIa After Inadequate Haemostasis in Complex Cardiac Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2005/02047
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Myocardial Ischemia; Blood Coagulation Disorders; Coronary Artery Disease; Heart Valve Diseases
Keywords: Cardiac surgical procedures; Surgical blood loss; Surgical haemostasis; Factor VIIa; Anaesthesia
MeSH Terms: conditions — Myocardial Ischemia; Blood Coagulation Disorders; Coronary Artery Disease; Heart Valve Diseases; Blood Loss, Surgical

INTERVENTIONS:
Drug: Recombinant Activated Factor VII

SUMMARY:
Aims and Hypotheses:

This randomised placebo controlled study will test the hypothesis that Recombinant Activated Factor VII (rVIIa) will improve haemostasis after an inadequate response to conventional therapy in complex cardiac surgery.

Major bleeding is still of concern in complex cardiac surgery. It has been shown to be associated with poorer patient outcome and results in the consumption of resources (hospital costs, manpower and blood bank reserves). This study has the potential to provide evidence that rVIIa can reduce transfusion requirements and improve patient outcome in a problematic aspect of complicated cardiac surgery.

The objective is to conduct a multi-centre randomised placebo controlled study that has been designed to scientifically evaluate the treatment of post bypass coagulopathy in the association with complex cardiac surgery. The trial design is based on clinical practice that has evolved over 2 years at the Austin Hospital during which 38 patients have received open label administration of rVIIa. There is currently no published RCT in this area and there is no TGA approval for the use of rVIIa for this indication.

DETAILED DESCRIPTION:
11. 3 Methods

Synopsis of Study:

A multicentred randomised, double blind, placebo-controlled trial evaluating the efficacy and safety of activated recombinant factor VII (rVIIa) in complex cardiac surgery.

Study will be conducted at Austin Hospital, Alfred Hospital and Warringal Private Hospital.

The study will have two arms:

1. Those who have inadequate haemostasis after initial standardised administration of coagulation factors and receive rVIIa. (Active arm)
2. Those who have inadequate haemostasis after initial standardised administration of coagulation factors and receive placebo. (Placebo arm)

   We anticipate from our preliminary series that 50% of enrolled subjects will achieve haemostasis after the initial standardised dose of coagulation factors and therefore don't receive trial medication. Identical data will be collected and will form an observational subgroup for analysis.

   The protocol allows for open label administration of rVIIa if adequate haemostasis is not achieved after two standardised administrations of coagulation factors and the trial medication. This would be within 2 hours of the completion of the first administration

   Primary endpoint will be "adequate haemostasis to enable chest closure" after administration of trial medication without the need for further intervention to improve coagulation.

   Secondary Endpoints, percentage of cases that haemostasis after first administration of coagulation factors alone Assessment of surgical field after administration of trial medication Time to closure of chest after administration of trial medication Transfusion requirements in post bypass period in theatre Transfusion requirements in ICU first 12 hours Mediastinal drainage in ICU first 12 hours Coagulation study results at various sample times Requirement for chest re-exploration Ventilation duration in ICU Duration of stay in ICU

   Inclusion Criteria:

   Patients with scheduled cardiac surgery undergoing the following procedures Double valve replacements or repair. Major thoracic aortic surgery including hypothermic circulatory arrest or descending aortic reconstruction.

   Valve repair or replacement in the setting of endocarditis Complex procedures requiring cardiopulmonary bypass duration anticipated to exceed 180 minutes in patients aged ³70 years

   Exclusion Criteria:

   Patient unable to give informed consent Patient refusal Allergy to rVIIa Allergy to aprotinin or prior exposure within 6 months Pre-existing congenital coagulopathy Pre-existing hypercoagulable state Patients in inclusion criteria whose actual bypass time does not exceed 180 minutes Unresolved surgical bleeding

   Withdrawal from Trial:

   At the discretion of treating physicians if the proposed transfusion protocol post CPB is inadequate to keep up with blood loss a patient can be withdrawn from the trial. Transfusion therapy according to current medical practice at the discretion of treating physicians will follow. rVIIa as per current hospital guidelines will be available. Data will still be collected in this group.

   Randomization Pharmacy will randomise patient after notified of entry into study. Blinded packaged trial medication will be sent to theatre.

   Surgical management Surgical technique will be at the discretion of treating surgeon but techniques that may affect haemostasis (eg. Use of biologic glues etc) will be recorded.

   Anaesthetic management Choice of anaesthetic agents will be at the discretion of treating anaesthetist.

   All patients will receive aprotinin 2 x 106 IV over 1 hour after test dose of 10,000 units over 5 minutes and 2 x 106 IV in the CPB circuit prime. 0.75 x 106 IV to infusion per hour.

   All patients will be haemofiltered on bypass.

   Core temperature monitoring on all patients. Standard technique to preserve patient temperature. Topical head cooling will be used if hypothermic circulatory arrest is needed.

   Cardiopulmonary bypass management

   Standardised CPB prime and circuits Cell saver for all patients Cardiotomy return for all patients

   Haemoglobin maintained between 6-8gm/dL during bypass. Aim for haemoglobin of 10gm/dL at time of weaning from bypass. Units of packed cells transfused on bypass will be recorded.

   Adequate rewarming core temp > 35° for 20 minutes.

   Alpha stat pH management. Acid-base pH 7.3-7.5, BE +/- 3 prior to weaning from bypass.

   Post bypass period

   Transfusion and trial medication administration guidelines are found on Flow Chart.

   Red Cell Transfusion Trigger Aim for haemoglobin concentration between 80 and 100 grams/litre using either banked or washed red cells.

   The planned "conventional therapy " of aprotinin and an initial administration predominately platelets (10 units), cryoprecipitate 3 mls/kg (high concentration of fibrinogen) and a moderate dose of fresh frozen plasma 5ml/kg is appropriate based on both our clinical experience and advice from the Australian Red Cross.

   If at anytime adherence to protocol at the discretion of treating medical staff is considered to place the patient at risk of inadequate transfusion, the patient can be withdrawn and transfusion commenced as determined by medical staff. Data will still be collected for these patients.

   The duration of protocol during transfusion is two hours. Either adequate haemostasis will have been achieved by the interventions as indicated in the protocol or the scenario of inadequate haemostasis despite two administrations of standardising coagulation factor and trial medications followed by open label administration of rVIIa will have evolved. If this is the case, ongoing transfusion, surgical and medical management will be at the discretion of medical staff. Administration of rVIIa can be considered after discussion with trial investigators. Data will still be collected for such patients.

   ICU Management Blood loss measurement in the closed drainage system must be documented at least once hourly, or more frequently if blood loss is excessive. The patient should be sat up in bed on arrival in ICU (this will allow CXR to be taken), before starting to measure drainage. On arrival to ICU coagulation studies should be performed and repeated 4 hours and 12 hours post arrival. .

   Postoperative transfusion according to established ICU protocol Blood loss > 250mL/hr NOTIFY SURGEON (CONSIDER RETURN TO THEATRE)

   CONSISTANT WITH CURRENT PRACTICE: - NO ADMINISTRATION OF rVIIa IN ICU

   Re-exploration for bleeding Any patient returning to theatre will be treated at the discretion of medical staff involved. The administration of rVIIa can be considered according to current guidelines. Administration of coagulation products at discretion of treating doctors.

   Randomisation will be co-ordinated and supervised by the Trial Pharmacy at the Austin Hospital.

   Due to the expense of the drug, instability in solution and the lack of availability of a similarly packaged placebo, the mechanism to "blind" medical staff in theatre will involve an independent registered nurse preparing the drug in an opaque syringe according to a sealed envelope indicating placebo or trial drug. Randomisation will be site specific for both the Austin Hospital and Warringal Private Hospital.

   Pharmacy will be notified when consent is obtained for a patient. Two doses or rVIIa will need to be sent to theatre. This will be stored in the blood fridge. Any unused drug will be returned to Pharmacy with full documentation of drug handling. Nursing staff involved in trial medication preparation will be educated regarding the necessity of not revealing whether actual drug or placebo was used.

   Statistics

   Power Analysis Based on our pilot data we anticipate 80% or more of the group receiving rVIIa will achieve haemostasis adequate for chest closure without any further intervention to improve coagulation. (Our primary endpoint) We conservatively estimate that only 30% or less of placebo group will achieve haemostasis adequate for chest closure without any further intervention to improve coagulation. Assuming a p value of < 0.5 and power of 0.8 analysis indicates that to show a 50% difference between groups 34 subjects are needed (17 in each arm). To allow for any withdrawals we plan to enrol 40 patients in the study. Based on current drug usage, the recruitment will take 2 years.

   Results Analysis Primary endpoints will be assessed by chi-squared analysis. Secondary endpoints parametric and non-parametric analysis as appropriate. No interim analysis is planned. Subgroup analysis according to procedure and surgeon will be performed.

   Bias Because of the small number of subjects in this trial, bias may be a problem. Unequal distribution of each of the four procedures may occur and influence results. The trial drug is thought to treat coagulopathic bleeding. Any superimposed surgical bleeding may cause bias.

   Adverse Events Patients undergoing cardiac surgery represent a population at relatively high risk of a range of perioperative complications inherent to their underlying disease, co-morbidities and the nature of the surgery being undertaken. In the pilot study the mortality rate was 25 %. It is not intended to report the occurrence all of these events to the Human Research and Ethics Committee. Any adverse events that do arise specifically in relation to the conduct of the proposed study will be reported to the Committee

   Feasibility Our pilot series of 40 cases from 2 centres was collected over a 24-month period. Assuming similar workloads and the addition of another centre ( Alfred Hospital) recruitment should be completed in 24 months.

   HREC approval has been granted by Austin Health for the Austin site. The same HREC is considering approval for the Warringal Private Hospital site, and the Alfred hospital will be seeking similar approval from its own HREC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scheduled cardiac surgery undergoing the following procedures
* Double valve replacements or repair.
* Major thoracic aortic surgery including hypothermic circulatory arrest or descending aortic reconstruction.
* Valve repair or replacement in the setting of endocarditis
* Complex procedures requiring cardiopulmonary bypass duration anticipated to exceed 180 minutes in patients aged ³70 years

Exclusion Criteria:

* Patient unable to give informed consent
* Patient refusal
* Allergy to rVIIa
* Allergy to aprotinin or prior exposure within 6 months
* Pre-existing congenital coagulopathy
* Pre-existing hypercoagulable state
* Patients in inclusion criteria whose actual bypass time does not exceed 180 minutes
* Unresolved surgical bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-06; Study Completion 2008-06

PRIMARY OUTCOMES:
Adequate haemostasis to enable chest closure after administration of trial medication without the need for further intervention to improve coagulation.

SECONDARY OUTCOMES:
Percentage of cases that haemostasis after first administration of coagulation factors alone
Assessment of surgical field after administration of trial medication
Time to closure of chest after administration of trial medication
Transfusion requirements in post bypass period in theatre
Transfusion requirements in ICU first 12 hours
Mediastinal drainage in ICU first 12 hours
Coagulation study results at various sample times
Requirement for chest re-exploration
Ventilation duration in ICU
Duration of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCall, FANZCA, Principal Investigator — Staff Anaesthetist
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Hedner U, Erhardtsen E. Potential role for rFVIIa in transfusion medicine. Transfusion. 2002 Jan;42(1):114-24. doi: 10.1046/j.1537-2995.2002.00017.x. No abstract available. PMID 11896322